CLINICAL TRIAL: NCT00453479
Title: A Randomised, Double-blind, Placebo-controlled, Dose Ascending, 2-cohort, Parallel Group Study to Examine the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Twice-daily Inhaled Doses of GSK233705B Formulated With the Excipient Magnesium Stearate in COPD Subjects for 7-days.
Brief Title: A Dose Ascending, Study To Examine The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of GSK233705B.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Diagnostic
Other Study IDs: AC2108378
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Results first posted 2018-02-08 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: muscarinic receptor,; bronchodilators; Chronic obstructive pulmonary disease,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK233705B

SUMMARY:
GSK233705 is a high-affinity specific muscarinic receptor (mAChR) antagonist which is being developed for the treatment of chronic obstructive pulmonary disease. This is a randomised, double-blind, placebo-controlled, dose ascending, parallel group study to examine the safety, tolerability, pharmacokinetics and pharmacodynamics of twice daily inhaled doses of GSK233705B for 7 days, in COPD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are between 40 and 75 years of age
* Female subjects must be of non-childbearing
* Subject diagnosed with COPD
* Body Mass Index 18.0 - 32.0 kg/m2 (inclusive)
* Subject is a smoker or an ex-smoker
* Subject has post-bronchodilator (200µg salbutamol) FEV1 of = 40% to = 80% of predicted normal.
* Subject has FEV1/FVC < 0.7 post-bronchodilator (200µg salbutamol).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Subject is available to complete all study measurements and procedures.
* Subjects have a 24hour holter recording that is within normal limits and does not demonstrate any clinically important abnormality that, in the opinion of the investigator, would make the subject unsuitable for participation in the study.

Exclusion Criteria:

* Subjects who have a past or present disease, which as judged by the Investigator and the Medical Monitor, may affect the outcome of this study.
* The subject has a positive pre-study alcohol screen.
* The subject has a positive pre-study drug screen.
* History of alcohol/drug abuse or dependence within 12 months of the study: Abuse
* The subject has a positive pregnancy test.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Subject has tested positive for HIV
* The subject has participated in a clinical trial and has received a drug or a new chemical entity within 60 days or 5 half-lives
* Exposure to more than three new chemical entities (NCE) within 10 months prior to the first dosing day or one NCE within 3 months prior to the first dosing day.
* The subject has donated a unit (400ml) of blood within 60 days of screening, or, intends to donate during the study.
* The subject has a known allergy or hypersensitivity to ipratropium bromide, atropine and any of its derivatives or milk protein/lactose.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the physician responsible, contraindicates their participation
* Subject has prostate hypertrophy or narrow angle glaucoma

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-03-28 (Actual); Primary Completion 2007-10-11 (Actual); Study Completion 2007-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Netherlands (4):
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Harderwijk
  - GSK Investigational Site, Utrecht
  - GSK Investigational Site, Zuidlaren

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: AC2108378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AC2108378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: AC2108378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AC2108378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AC2108378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AC2108378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AC2108378 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 29 March 2007 to 11 October 2007, total of 23 participants with chronic obstructive pulmonary disease (COPD) were randomized at four centres in the Netherlands. DISKUS™ is registered product of GlaxoSmithKline.
Groups:
- Placebo: Participants entered into Cohort I received single inhaled dose of dry powder inhaler (DPI) of matching placebo administered twice daily for 7 days and those in Cohort II received two inhaled dose of DPI matching placebo administered twice daily for 7 days. Matching placebo was administered via the DISKUS inhaler (60 doses) and was formulated with lactose only as a vehicle to make 12.5 milligrams (mg).
- GSK233705 50 µg Twice Daily: Participants entered into Cohort I received single inhaled dose of DPI of GSK233705 50 micrograms (µg) administered twice daily for 7 days. GSK233705 50 μg blister was administered via the DISKUS inhaler (60 doses) and was formulated with magnesium stearate (0.5%) as a vehicle to make 12.5 mg.
- GSK233705 100 µg Twice Daily: Participants entered into Cohort II received two inhaled dose of DPI GSK233705 (50 µg) administered twice daily for 7 days. GSK233705 50 μg blister was administered via the DISKUS inhaler (60 doses) and was formulated with magnesium stearate (0.5%) as a vehicle to make 12.5 mg.
Period: Overall Study
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Started | 6 | 9 | 8
Completed | 6 | 9 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants entered into Cohort I received single inhaled dose of DPI of matching placebo administered twice daily for 7 days and those in Cohort II received two inhaled dose of DPI matching placebo administered twice daily for 7 days. Matching placebo was administered via the DISKUS inhaler (60 doses) formulated with lactose only as a vehicle to make 12.5 mg.
- GSK233705 50 µg Twice Daily: Participants entered into Cohort I received single inhaled dose of DPI of GSK233705 50 µg administered twice daily for 7 days. GSK233705 50 μg blister was administered via the DISKUS inhaler (60 doses) and was formulated with magnesium stearate (0.5%) as a vehicle to make 12.5 mg.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily | Total
Number analyzed (Participants) | 6 | 9 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.0 (11.15) | 66.4 (6.31) | 59.0 (7.27) | 62.2 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 4
  Male | 5 | 9 | 5 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 9 | 8 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) and Serious Adverse Events (SAE)
Description: An AE was defined as any untoward medical occurrence (MO) in a participant temporally associated with the use of a medicinal product (MP), whether or not considered related to the MP and can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with its use. The SAE was any untoward MO that, at any dose, results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect, that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition.
Time Frame: Up to follow-up (approximately 45 days)
Population: All subject population included all available data on participants who had received at least one dose of study medication (including placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Participants
  Any AE | 4 | 4 | 4
  Any SAE | 0 | 0 | 0

2. Primary Outcome: Summary of Mean Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured subsequent to 12 lead electrocardiogram (ECG). Baseline was defined as the mean of the three planned pre-dose measurements. It was assessed on Baseline (triplicate), 15, 30 minutes, 1.5, 4, 8 and 24 hours on Day 1 and 7.
Time Frame: Up to Day 7 (24 hours post-dose)
Population: All subject population was used.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Millimeters of mercury
  SBP, Day 1, Baseline | 129.2 (15.37) | 127.7 (9.03) | 129.6 (11.78)
  SBP, Day 1, 15 minutes | 130.0 (12.84) | 130.0 (8.99) | 130.6 (16.04)
  SBP, Day 1, 30 minutes | 126.0 (14.24) | 123.7 (10.85) | 128.4 (9.32)
  SBP, Day 1, 1.5 hour | 131.2 (16.17) | 124.1 (13.01) | 133.5 (18.47)
  SBP, Day 1, 4 hour | 126.2 (17.52) | 124.8 (9.90) | 132.1 (12.96)
  SBP, Day 1, 8 hour | 132.8 (14.26) | 121.1 (9.44) | 124.0 (13.03)
  SBP, Day 1, 24 hour | 131.5 (13.49) | 123.1 (7.64) | 129.6 (16.10)
  SBP, Day 7, Baseline | 124.6 (15.25) | 122.7 (11.94) | 123.9 (9.21)
  SBP, Day 7, 15 minutes | 127.5 (16.43) | 123.1 (12.75) | 123.6 (11.13)
  SBP, Day 7, 30 minutes | 122.5 (22.21) | 124.6 (13.41) | 119.5 (9.58)
  SBP, Day 7, 1.5 hour | 127.0 (16.12) | 122.8 (12.55) | 123.9 (10.86)
  SBP, Day 7, 4 hour | 127.2 (13.26) | 122.7 (10.78) | 123.9 (15.42)
  SBP, Day 7, 8 hour | 131.0 (20.71) | 123.3 (12.59) | 123.1 (13.22)
  SBP, Day 7, 24 hour | 130.3 (15.96) | 126.6 (11.67) | 129.1 (10.64)
  DBP, Day 1, Baseline | 74.7 (8.69) | 77.4 (4.29) | 80.0 (10.60)
  DBP, Day 1, 15 minutes | 78.0 (7.43) | 78.9 (4.11) | 81.1 (9.95)
  DBP, Day 1, 30 minutes | 76.2 (8.80) | 77.0 (5.00) | 77.3 (10.61)
  DBP, Day 1, 1.5 hour | 74.8 (6.82) | 76.2 (4.02) | 78.4 (8.35)
  DBP, Day 1, 4 hour | 77.3 (9.42) | 80.3 (5.32) | 77.9 (12.08)
  DBP, Day 1, 8 hour | 75.3 (9.16) | 75.7 (5.41) | 72.6 (10.95)
  DBP, Day 1, 24 hour | 77.2 (6.05) | 77.4 (3.32) | 76.0 (12.98)
  DBP, Day 7, Baseline | 77.0 (8.80) | 76.7 (5.15) | 75.4 (7.21)
  DBP, Day 7, 15 minutes | 82.5 (10.97) | 76.1 (4.65) | 75.0 (9.97)
  DBP, Day 7, 30 minutes | 78.8 (10.70) | 77.7 (4.58) | 74.9 (11.13)
  DBP, Day 7, 1.5 hour | 78.2 (10.57) | 76.8 (4.27) | 73.6 (8.99)
  DBP, Day 7, 4 hour | 79.3 (7.69) | 78.2 (4.55) | 74.0 (12.72)
  DBP, Day 7, 8 hour | 79.0 (12.66) | 75.6 (5.15) | 73.4 (8.33)
  DBP, Day 7, 24 hour | 78.8 (9.39) | 77.4 (4.61) | 73.4 (11.50)

3. Primary Outcome: Summary of Mean Heart Rate
Description: Heart rate was measured subsequent to 12 lead ECG. Baseline was defined as the mean of the three planned pre-dose measurements. It was assessed on Baseline (triplicate), 15, 30 minutes, 1.5, 4, 8 and 24 hours on Day 1 and 7.
Time Frame: Up to Day 7 (24 hour post dose)
Population: All subject population was used.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Beats per minute
  Day 1, Baseline | 65.7 (7.07) | 66.7 (9.68) | 71.5 (8.50)
  Day 1, 15 minutes | 62.2 (8.06) | 65.1 (8.07) | 70.4 (10.57)
  Day 1, 30 minutes | 61.2 (5.78) | 64.9 (8.57) | 66.6 (7.42)
  Day 1, 1.5 hour | 64.7 (9.52) | 62.7 (9.63) | 64.9 (6.29)
  Day 1, 4 hour | 63.2 (6.31) | 66.6 (14.57) | 64.0 (8.37)
  Day 1, 8 hour | 65.7 (5.75) | 68.1 (11.12) | 66.9 (6.01)
  Day 1, 24 hour | 62.3 (10.25) | 68.1 (13.13) | 65.5 (8.45)
  Day 7, Baseline | 63.6 (4.62) | 67.0 (8.20) | 67.8 (8.30)
  Day 7, 15 minutes | 65.3 (6.56) | 68.3 (14.27) | 64.5 (6.55)
  Day 7, 30 minutes | 63.3 (6.25) | 66.7 (11.79) | 65.0 (7.33)
  Day 7, 1.5 hour | 60.0 (7.01) | 64.0 (11.61) | 62.5 (8.25)
  Day 7, 4 hour | 64.3 (8.91) | 66.2 (12.72) | 63.0 (8.43)
  Day 7, 8 hour | 65.3 (4.89) | 66.1 (7.62) | 66.3 (5.47)
  Day 7, 24 hour | 68.0 (9.78) | 70.2 (17.22) | 65.5 (5.98)

4. Primary Outcome: Maximum Value of SBP and DBP (0-4 Hour) for the Morning Dose
Description: Blood pressure was measured subsequent to 12 lead ECG. Baseline was defined as the mean of the three planned pre-dose measurements. It was assessed on pre-dose, 15, 30 minutes, 1.5 and 4 hours on Day 1 and 7. Data for adjusted mean is presented as least square mean.
Time Frame: Up to Day 7 (0-4 hour)
Population: All subject population
Measure: Least Squares Mean (95% Confidence Interval); unit: Millimeters of mercury
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Millimeters of mercury
  SBP, Day 1 | 132.52 [123.46 to 141.58] | 131.56 [124.15 to 138.97] | 138.73 [130.88 to 146.59]
  SBP, Day 7 | 132.43 [125.61 to 139.26] | 128.33 [122.75 to 133.92] | 127.67 [121.76 to 133.59]
  DBP, Day 1 | 81.21 [77.72 to 84.71] | 81.80 [79.00 to 84.60] | 82.19 [79.17 to 85.22]
  DBP, Day 7 | 86.14 [82.24 to 90.03] | 79.50 [76.38 to 82.62] | 75.33 [71.96 to 78.70]
Statistical Analysis 1: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -0.97, 95% CI 2-sided [-12.68 to 10.75], Standard Error of Mean 5.596 — Comparison of SBP Day 1
Statistical Analysis 2: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -4.10, 95% CI 2-sided [-12.92 to 4.72], Standard Error of Mean 4.215 — Comparison of SBP Day 7
Statistical Analysis 3: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 6.21, 95% CI 2-sided [-5.78 to 18.19], Standard Error of Mean 5.727 — Comparison of SBP Day 1
Statistical Analysis 4: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -4.76, 95% CI 2-sided [-13.79 to 4.27], Standard Error of Mean 4.314 — Comparison of SBP Day 7
Statistical Analysis 5: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.58, 95% CI 2-sided [-3.89 to 5.06], Standard Error of Mean 2.138 — Comparison of DBP Day 1
Statistical Analysis 6: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -6.64, 95% CI 2-sided [-11.62 to -1.65], Standard Error of Mean 2.382 — Comparison of DBP Day 7
Statistical Analysis 7: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.98, 95% CI 2-sided [-3.73 to 5.68], Standard Error of Mean 2.248 — Comparison of DBP Day 1
Statistical Analysis 8: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -10.81, 95% CI 2-sided [-16.05 to -5.57], Standard Error of Mean 2.504 — Comparison of DBP Day 7

5. Primary Outcome: Maximum Value of Heart Rate (0-4 Hour) for the Morning Dose
Description: Heart rate was measured subsequent to 12 lead ECG. Baseline was defined as the mean of the three planned pre-dose measurements. It was assessed on pre-dose, 15, 30 minutes, 1.5 and 4 hours on Day 1 and 7. Data for adjusted mean is presented as least square mean.
Time Frame: Up to Day 7 (0-4 hour)
Population: All subject population was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Beats per minute
  Day 1 | 68.32 [62.19 to 74.46] | 70.58 [65.60 to 75.57] | 68.48 [63.07 to 73.89]
  Day 7 | 69.30 [63.10 to 75.50] | 71.92 [66.89 to 76.96] | 63.86 [58.39 to 69.33]
Statistical Analysis 1: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 2.26, 95% CI 2-sided [-5.58 to 10.10], Standard Error of Mean 3.745 — Comparison at Day 1
Statistical Analysis 2: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 2.62, 95% CI 2-sided [-5.30 to 10.54], Standard Error of Mean 3.785 — Comparison at Day 7
Statistical Analysis 3: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.16, 95% CI 2-sided [-8.17 to 8.48], Standard Error of Mean 3.979 — Comparison at Day 1
Statistical Analysis 4: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -5.44, 95% CI 2-sided [-13.86 to 2.97], Standard Error of Mean 4.021 — Comparison at Day 7

6. Primary Outcome: Weighted Mean of SBP and DBP (0-4 Hour) for the Morning Dose
Description: as for outcome 4
Time Frame: Up to Day 7 (0-4 hour)
Population: All subject population was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: Millimeters of mercury
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Millimeters of mercury
  SBP, Day 1 | 128.31 [120.84 to 135.77] | 125.53 [119.43 to 131.64] | 131.32 [124.85 to 137.79]
  SBP, Day 7 | 125.87 [119.53 to 132.21] | 123.99 [118.81 to 129.17] | 122.37 [116.88 to 127.87]
  DBP, Day 1 | 78.22 [75.24 to 81.20] | 77.94 [75.56 to 80.33] | 76.47 [73.89 to 79.04]
  DBP, Day 7 | 81.37 [77.91 to 84.84] | 77.49 [74.71 to 80.26] | 71.99 [68.99 to 74.98]
Statistical Analysis 1: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -2.78, 95% CI 2-sided [-12.43 to 6.87], Standard Error of Mean 4.611 — Comparison of SBP Day 1
Statistical Analysis 2: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -1.88, 95% CI 2-sided [-10.07 to 6.31], Standard Error of Mean 3.913 — Comparison of SBP Day 7
Statistical Analysis 3: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 3.01, 95% CI 2-sided [-6.87 to 12.88], Standard Error of Mean 4.718 — Comparison of SBP Day 1
Statistical Analysis 4: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -3.50, 95% CI 2-sided [-11.88 to 4.89], Standard Error of Mean 4.005 — Comparison of SBP Day 7
Statistical Analysis 5: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -0.28, 95% CI 2-sided [-4.09 to 3.54], Standard Error of Mean 1.822 — Comparison of DBP Day 1
Statistical Analysis 6: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -3.89, 95% CI 2-sided [-8.32 to 0.54], Standard Error of Mean 2.116 — Comparison of DBP Day 7
Statistical Analysis 7: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -1.75, 95% CI 2-sided [-5.76 to 2.26], Standard Error of Mean 1.916 — Comparison of DBP Day 1
Statistical Analysis 8: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -9.39, 95% CI 2-sided [-14.04 to -4.73], Standard Error of Mean 2.224 — Comparison of DBP Day 7

7. Primary Outcome: Weighted Mean of Heart Rate (0-4 Hour) for the Morning Dose
Description: as for outcome 5
Time Frame: Up to Day 7 (0-4 hour)
Population: All subject population was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Beats per minute
  Day 1 | 65.46 [61.04 to 69.88] | 65.60 [62.00 to 69.19] | 62.79 [58.89 to 66.70]
  Day 7 | 64.31 [59.70 to 68.92] | 66.70 [62.96 to 70.44] | 60.47 [56.40 to 64.53]
Statistical Analysis 1: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.14, 95% CI 2-sided [-5.52 to 5.79], Standard Error of Mean 2.700 — Comparison at Day 1
Statistical Analysis 2: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 2.39, 95% CI 2-sided [-3.50 to 8.28], Standard Error of Mean 2.813 — Comparison at Day 7
Statistical Analysis 3: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -2.67, 95% CI 2-sided [-8.67 to 3.34], Standard Error of Mean 2.869 — Comparison at Day 1
Statistical Analysis 4: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -3.84, 95% CI 2-sided [-10.10 to 2.41], Standard Error of Mean 2.989 — Comparison at Day 7

8. Primary Outcome: Number of Participants With Abnormal 12-lead ECG Findings
Description: Single measurements were taken at all time points. The pre-dose values were classed as Baseline. Data for number of participants with normal, abnormal not clinically significant and abnormal clinically significant is presented. It was assessed on Baseline (triplicate), 15, 30 minutes, 1.5, 4, 8 and 24 hours on Day 1 and 7.
Time Frame: Up to Day 7 (24 hour post dose)
Population: All subject population was used. Only those participants available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Participants
  Day 1, Baseline: Normal | 3 | 5 | 6
  Day 1, Baseline: Abnormal not clinically significant | 3 | 4 | 2
  Day 1, Baseline: Abnormal clinically significant | 0 | 0 | 0
  Day 1, 15 minutes: Normal | 2 | 4 | 5
  Day 1, 15 minutes: Abnormal not clinically significant | 4 | 5 | 3
  Day 1, 15 minutes: Abnormal clinically significant | 0 | 0 | 0
  Day 1, 30 minutes: Normal | 3 | 5 | 5
  Day 1, 30 minutes: Abnormal not clinically significant | 3 | 4 | 3
  Day 1, 30 minutes: Abnormal clinically significant | 0 | 0 | 0
  Day 1, 1.5 hour: Normal | 3 | 7 | 3
  Day 1, 1.5 hour: Abnormal not clinically significant | 3 | 2 | 5
  Day 1, 1.5 hour: Abnormal clinically significant | 0 | 0 | 0
  Day 1, 4 hour: Normal | 2 | 3 | 5
  Day 1, 4 hour: Abnormal not clinically significant | 4 | 6 | 3
  Day 1, 4 hour: Abnormal clinically significant | 0 | 0 | 0
  Day 1, 8 hour: Normal | 3 | 5 | 5
  Day 1, 8 hour: Abnormal not clinically significant | 3 | 4 | 3
  Day 1, 8 hour: Abnormal clinically significant | 0 | 0 | 0
  Day 1, 24 hour: Normal | 3 | 5 | 5
  Day 1, 24 hour: Abnormal not clinically significant | 3 | 4 | 3
  Day 1, 24 hour: Abnormal clinically significant | 0 | 0 | 0
  Day 7, Baseline: Normal | 3 | 5 | 6
  Day 7, Baseline: Abnormal not clinically significant | 3 | 4 | 2
  Day 7, Baseline: Abnormal clinically significant | 0 | 0 | 0
  Day 7, 15 minutes: Normal | 2 | 4 | 6
  Day 7, 15 minutes: Abnormal not clinically significant | 4 | 5 | 2
  Day 7, 15 minutes: Abnormal clinically significant | 0 | 0 | 0
  Day 7, 30 minutes: Normal | 2 | 5 | 6
  Day 7, 30 minutes: Abnormal not clinically significant | 4 | 4 | 2
  Day 7, 30 minutes: Abnormal clinically significant | 0 | 0 | 0
  Day 7, 1.5 hour: Normal | 2 | 3 | 6
  Day 7, 1.5 hour: Abnormal not clinically significant | 4 | 6 | 2
  Day 7, 1.5 hour: Abnormal clinically significant | 0 | 0 | 0
  Day 7, 4 hour: number analyzed (Participants) | 5 | 9 | 8
  Day 7, 4 hour: Normal | 1 | 5 | 6
  Day 7, 4 hour: Abnormal not clinically significant | 4 | 4 | 2
  Day 7, 4 hour: Abnormal clinically significant | 0 | 0 | 0
  Day 7, 8 hour: Normal | 3 | 5 | 6
  Day 7, 8 hour: Abnormal not clinically significant | 3 | 4 | 2
  Day 7, 8 hour: Abnormal clinically significant | 0 | 0 | 0
  Day 7, 24 hour: Normal | 2 | 4 | 6
  Day 7, 24 hour: Abnormal not clinically significant | 4 | 5 | 2
  Day 7, 24 hour: Abnormal clinically significant | 0 | 0 | 0

9. Primary Outcome: Maximum Value (0-4 Hour) for the Morning Dose of ECG Parameters Corrected According to Fredericia's Formula (QTcF) and Corrected According to Bazett's Formula (QTc B)
Description: Baseline was defined as the mean of the three planned pre-dose measurements. It was assessed on pre-dose, 15, 30 minutes, 1.5 and 4 hours on Day 1 and 7. Data for adjusted mean is presented as least square mean.
Time Frame: Up to Day 7 (0-4 hour)
Population: All subject population was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: Milliseconds
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Milliseconds
  QTcB, Day 1 | 406.29 [392.99 to 419.60] | 410.71 [399.93 to 421.48] | 416.86 [405.30 to 428.42]
  QTcB, Day 7 | 400.21 [389.18 to 411.23] | 409.23 [400.30 to 418.16] | 416.71 [407.13 to 426.29]
  QTcF, Day 1 | 402.97 [388.50 to 417.43] | 405.10 [393.37 to 416.83] | 420.63 [408.14 to 433.11]
  QTcF, Day 7 | 395.77 [387.16 to 404.37] | 408.06 [401.08 to 415.04] | 418.08 [410.66 to 425.51]
Statistical Analysis 1: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 4.42, 95% CI 2-sided [-12.66 to 21.49], Standard Error of Mean 8.157 — Comparison of QTcB Day 1
Statistical Analysis 2: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 9.02, 95% CI 2-sided [-5.13 to 23.17], Standard Error of Mean 6.760 — Comparison of QTcB Day 7
Statistical Analysis 3: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 10.57, 95% CI 2-sided [-7.24 to 28.38], Standard Error of Mean 8.510 — Comparison of QTcB Day 1
Statistical Analysis 4: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 16.50, 95% CI 2-sided [1.74 to 31.26], Standard Error of Mean 7.052 — Comparison of QTcB Day 7
Statistical Analysis 5: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 2.13, 95% CI 2-sided [-16.51 to 20.78], Standard Error of Mean 8.908 — Comparison of QTcF Day 1
Statistical Analysis 6: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 12.29, 95% CI 2-sided [1.20 to 23.38], Standard Error of Mean 5.298 — Comparison of QTcF Day 7
Statistical Analysis 7: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 17.66, 95% CI 2-sided [-1.53 to 36.85], Standard Error of Mean 9.171 — Comparison of QTcF Day 1
Statistical Analysis 8: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 22.32, 95% CI 2-sided [10.90 to 33.73], Standard Error of Mean 5.454 — Comparison of QTcF Day 7

10. Primary Outcome: Weighted Mean (0-4 h) for the Morning Dose of ECG Parameters QTcF and QTc B
Description: as for outcome 9
Time Frame: Up to Day 7 (0-4 hour)
Population: All subject population was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: Milliseconds
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Milliseconds
  QTcB, Day 1 | 393.77 [385.19 to 402.36] | 403.33 [396.38 to 410.28] | 405.25 [397.79 to 412.71]
  QTcB, Day 7 | 392.54 [382.92 to 402.17] | 400.93 [393.14 to 408.73] | 407.83 [399.46 to 416.19]
  QTcF, Day 1 | 391.25 [383.74 to 398.75] | 399.57 [393.48 to 405.66] | 408.08 [401.60 to 414.56]
  QTcF, Day 7 | 390.72 [382.21 to 399.22] | 399.47 [392.57 to 406.37] | 411.18 [403.83 to 418.52]
Statistical Analysis 1: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 9.55, 95% CI 2-sided [-1.46 to 20.57], Standard Error of Mean 5.262 — Comparison of QTcB Day 1
Statistical Analysis 2: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 8.39, 95% CI 2-sided [-3.97 to 20.74], Standard Error of Mean 5.902 — Comparison of QTcB Day 7
Statistical Analysis 3: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 11.47, 95% CI 2-sided [-0.02 to 22.96], Standard Error of Mean 5.490 — Comparison of QTcB Day 1
Statistical Analysis 4: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 15.28, 95% CI 2-sided [2.39 to 28.17], Standard Error of Mean 6.157 — Comparison of QTcB Day 7
Statistical Analysis 5: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 8.32, 95% CI 2-sided [-1.35 to 18.00], Standard Error of Mean 4.622 — Comparison of QTcF Day 1
Statistical Analysis 6: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 8.75, 95% CI 2-sided [-2.21 to 19.72], Standard Error of Mean 5.239 — Comparison of QTcF Day 7
Statistical Analysis 7: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 16.83, 95% CI 2-sided [6.87 to 26.79], Standard Error of Mean 4.759 — Comparison of QTcF Day 1
Statistical Analysis 8: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 20.46, 95% CI 2-sided [9.17 to 31.75], Standard Error of Mean 5.394 — Comparison of QTcF Day 7

11. Primary Outcome: Summary of Mean Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC)
Description: It was assessed on 1, 2, 4, 9, 12 and 24 hours on Days 1 and 7. Also on Day 7, it was measured on 0 hour (Baseline). At all time points 3 measurements were taken and formal statistical analysis was carried out on the derived maximum readings. Data for adjusted mean is presented as least square mean.
Time Frame: Up to Day 7 (24-hour post dose)
Population: All subject population was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Liters
  FEV1, Day 1, 1 hour | 1.713 [1.571 to 1.855] | 1.860 [1.749 to 1.971] | 1.919 [1.799 to 2.039]
  FEV1, Day 1, 2 hour | 1.726 [1.581 to 1.871] | 1.897 [1.783 to 2.011] | 2.055 [1.931 to 2.178]
  FEV1, Day 1, 4 hour | 1.687 [1.556 to 1.818] | 1.747 [1.645 to 1.850] | 1.953 [1.842 to 2.064]
  FEV1, Day 1, 9 hour | 1.614 [1.430 to 1.798] | 1.764 [1.620 to 1.908] | 1.934 [1.778 to 2.090]
  FEV1, Day 1, 12 hour | 1.616 [1.445 to 1.786] | 1.740 [1.607 to 1.874] | 1.788 [1.643 to 1.932]
  FEV1, Day 1, 24 hour | 1.644 [1.456 to 1.832] | 1.807 [1.660 to 1.955] | 1.798 [1.638 to 1.957]
  FEV1, Day 7, Baseline | 1.515 [1.352 to 1.678] | 1.751 [1.623 to 1.879] | 1.771 [1.633 to 1.909]
  FEV1, Day 7, 1 hour | 1.560 [1.361 to 1.759] | 1.789 [1.633 to 1.945] | 1.856 [1.687 to 2.025]
  FEV1, Day 7, 2 hour | 1.665 [1.463 to 1.867] | 1.760 [1.602 to 1.918] | 1.867 [1.696 to 2.038]
  FEV1, Day 7, 4 hour | 1.604 [1.413 to 1.796] | 1.777 [1.627 to 1.927] | 1.811 [1.649 to 1.974]
  FEV1, Day 7, 9 hour | 1.598 [1.367 to 1.830] | 1.804 [1.623 to 1.985] | 1.878 [1.682 to 2.074]
  FEV1, Day 7, 12 hour | 1.526 [1.306 to 1.746] | 1.746 [1.573 to 1.919] | 1.719 [1.532 to 1.906]
  FEV1, Day 7, 24 hour | 1.614 [1.380 to 1.848] | 1.820 [1.636 to 2.004] | 1.793 [1.595 to 1.992]
  FVC, Day 1, 1 hour | 3.623 [3.312 to 3.935] | 3.761 [3.508 to 4.013] | 3.776 [3.506 to 4.045]
  FVC, Day 1, 2 hour | 3.689 [3.387 to 3.990] | 3.819 [3.575 to 4.063] | 4.009 [3.748 to 4.271]
  FVC, Day 1, 4 hour | 3.596 [3.303 to 3.889] | 3.558 [3.321 to 3.795] | 3.907 [3.653 to 4.161]
  FVC, Day 1, 9 hour | 3.571 [3.262 to 3.880] | 3.631 [3.381 to 3.881] | 3.919 [3.652 to 4.187]
  FVC, Day 1, 12 hour | 3.544 [3.188 to 3.900] | 3.658 [3.370 to 3.947] | 3.789 [3.480 to 4.097]
  FVC, Day 1, 24 hour | 3.593 [3.288 to 3.898] | 3.708 [3.461 to 3.955] | 3.755 [3.491 to 4.019]
  FVC, Day 7, Baseline | 3.266 [2.836 to 3.695] | 3.628 [3.280 to 3.976] | 3.801 [3.428 to 4.173]
  FVC, Day 7, 1 hour | 3.375 [2.962 to 3.789] | 3.644 [3.309 to 3.979] | 3.999 [3.640 to 4.357]
  FVC, Day 7, 2 hour | 3.503 [3.097 to 3.909] | 3.524 [3.195 to 3.853] | 3.962 [3.610 to 4.314]
  FVC, Day 7, 4 hour | 3.465 [3.065 to 3.865] | 3.642 [3.318 to 3.966] | 3.929 [3.583 to 4.275]
  FVC, Day 7, 9 hour | 3.449 [3.037 to 3.860] | 3.714 [3.381 to 4.048] | 3.894 [3.537 to 4.250]
  FVC, Day 7, 12 hour | 3.316 [2.868 to 3.765] | 3.683 [3.320 to 4.046] | 3.600 [3.212 to 3.989]
  FVC, Day 7, 24 hour | 3.449 [3.040 to 3.857] | 3.691 [3.360 to 4.022] | 3.832 [3.478 to 4.187]
Statistical Analysis 1: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.147, 95% CI 2-sided [-0.035 to 0.328], Standard Error of Mean 0.0921 — Comparison of FEV1, Day 1, 1 hour
Statistical Analysis 2: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.171, 95% CI 2-sided [-0.015 to 0.357], Standard Error of Mean 0.0944 — Comparison of FEV1, Day 1, 2 hour
Statistical Analysis 3: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.060, 95% CI 2-sided [-0.107 to 0.228], Standard Error of Mean 0.0850 — Comparison of FEV1, Day 1, 4 hour
Statistical Analysis 4: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.150, 95% CI 2-sided [-0.085 to 0.386], Standard Error of Mean 0.1195 — Comparison of FEV1, Day 1, 9 hour
Statistical Analysis 5: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.124, 95% CI 2-sided [-0.094 to 0.343], Standard Error of Mean 0.1107 — Comparison of FEV1, Day 1, 12 hour
Statistical Analysis 6: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.163, 95% CI 2-sided [-0.077 to 0.404], Standard Error of Mean 0.1220 — Comparison of FEV1, Day 1, 24 hour
Statistical Analysis 7: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.236, 95% CI 2-sided [0.027 to 0.444], Standard Error of Mean 0.1057 — Comparison of FEV1, Day 7, Baseline
Statistical Analysis 8: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.229, 95% CI 2-sided [-0.026 to 0.483], Standard Error of Mean 0.1292 — Comparison of FEV1, Day 7, 1 hour
Statistical Analysis 9: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.095, 95% CI 2-sided [-0.163 to 0.353], Standard Error of Mean 0.1309 — Comparison of FEV1, Day 7, 2 hour
Statistical Analysis 10: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.173, 95% CI 2-sided [-0.072 to 0.418], Standard Error of Mean 0.1243 — Comparison of FEV1, Day 7, 4 hour
Statistical Analysis 11: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.205, 95% CI 2-sided [-0.090 to 0.501], Standard Error of Mean 0.1499 — Comparison of FEV1, Day 7, 9 hour
Statistical Analysis 12: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.220, 95% CI 2-sided [-0.062 to 0.502], Standard Error of Mean 0.1430 — Comparison of FEV1, Day 7, 12 hour
Statistical Analysis 13: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.206, 95% CI 2-sided [-0.093 to 0.506], Standard Error of Mean 0.1520 — Comparison of FEV1, Day 7, 24 hour
Statistical Analysis 14: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.206, 95% CI 2-sided [0.015 to 0.397], Standard Error of Mean 0.0970 — Comparison of FEV1, Day 1, 1 hour
Statistical Analysis 15: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.329, 95% CI 2-sided [0.133 to 0.525], Standard Error of Mean 0.0994 — Comparison of FEV1, Day 1, 2 hour
Statistical Analysis 16: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.266, 95% CI 2-sided [0.090 to 0.443], Standard Error of Mean 0.0895 — Comparison of FEV1, Day 1, 4 hour
Statistical Analysis 17: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.320, 95% CI 2-sided [0.072 to 0.568], Standard Error of Mean 0.1258 — Comparison of FEV1, Day 1, 9 hour
Statistical Analysis 18: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.172, 95% CI 2-sided [-0.058 to 0.402], Standard Error of Mean 0.1165 — Comparison of FEV1, Day 1, 12 hour
Statistical Analysis 19: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.154, 95% CI 2-sided [-0.099 to 0.407], Standard Error of Mean 0.1285 — Comparison of FEV1, Day 1, 24 hour
Statistical Analysis 20: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.256, 95% CI 2-sided [0.036 to 0.475], Standard Error of Mean 0.1113 — Comparison of FEV1, Day 7, Baseline
Statistical Analysis 21: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.296, 95% CI 2-sided [0.027 to 0.564], Standard Error of Mean 0.1361 — Comparison of FEV1, Day 7, 1 hour
Statistical Analysis 22: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.202, 95% CI 2-sided [-0.069 to 0.474], Standard Error of Mean 0.1378 — Comparison of FEV1, Day 7, 2 hour
Statistical Analysis 23: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.207, 95% CI 2-sided [-0.051 to 0.465], Standard Error of Mean 0.1309 — Comparison of FEV1, Day 7, 4 hour
Statistical Analysis 24: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.280, 95% CI 2-sided [-0.032 to 0.591], Standard Error of Mean 0.1579 — Comparison of FEV1, Day 7, 9 hour
Statistical Analysis 25: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.193, 95% CI 2-sided [-0.104 to 0.490], Standard Error of Mean 0.1506 — Comparison of FEV1, Day 7, 12 hour
Statistical Analysis 26: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.180, 95% CI 2-sided [-0.136 to 0.495], Standard Error of Mean 0.1601 — Comparison of FEV1, Day 7, 24 hour
Statistical Analysis 27: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.137, 95% CI 2-sided [-0.263 to 0.537], Standard Error of Mean 0.2029 — Comparison of FVC, Day 1, 1 hour
Statistical Analysis 28: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.131, 95% CI 2-sided [-0.257 to 0.518], Standard Error of Mean 0.1965 — Comparison of FVC, Day 1, 2 hour
Statistical Analysis 29: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -0.038, 95% CI 2-sided [-0.414 to 0.338], Standard Error of Mean 0.1908 — Comparison of FVC, Day 1, 4 hour
Statistical Analysis 30: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.060, 95% CI 2-sided [-0.337 to 0.457], Standard Error of Mean 0.2013 — Comparison of FVC, Day 1, 9 hour
Statistical Analysis 31: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.115, 95% CI 2-sided [-0.343 to 0.572], Standard Error of Mean 0.2322 — Comparison of FVC, Day 1, 12 hour
Statistical Analysis 32: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.115, 95% CI 2-sided [-0.277 to 0.507], Standard Error of Mean 0.1988 — Comparison of FVC, Day 1, 24 hour
Statistical Analysis 33: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.362, 95% CI 2-sided [-0.190 to 0.914], Standard Error of Mean 0.2801 — Comparison of FVC, Day 7, Baseline
Statistical Analysis 34: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.269, 95% CI 2-sided [-0.263 to 0.800], Standard Error of Mean 0.2696 — Comparison of FVC, Day 7, 1 hour
Statistical Analysis 35: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.021, 95% CI 2-sided [-0.501 to 0.543], Standard Error of Mean 0.2648 — Comparison of FVC, Day 7, 2 hour
Statistical Analysis 36: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.177, 95% CI 2-sided [-0.337 to 0.691], Standard Error of Mean 0.2606 — Comparison of FVC, Day 7, 4 hour
Statistical Analysis 37: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.266, 95% CI 2-sided [-0.263 to 0.795], Standard Error of Mean 0.2684 — Comparison of FVC, Day 7, 9 hour
Statistical Analysis 38: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.367, 95% CI 2-sided [-0.209 to 0.943], Standard Error of Mean 0.2923 — Comparison of FVC, Day 7, 12 hour
Statistical Analysis 39: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.242, 95% CI 2-sided [-0.283 to 0.768], Standard Error of Mean 0.2665 — Comparison of FVC, Day 7, 24 hour
Statistical Analysis 40: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.152, 95% CI 2-sided [-0.263 to 0.567], Standard Error of Mean 0.2106 — Comparison of FVC, Day 1, 1 hour
Statistical Analysis 41: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.321, 95% CI 2-sided [-0.081 to 0.723], Standard Error of Mean 0.2039 — Comparison of FVC, Day 1, 2 hour
Statistical Analysis 42: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.311, 95% CI 2-sided [-0.079 to 0.701], Standard Error of Mean 0.1981 — Comparison of FVC, Day 1, 4 hour
Statistical Analysis 43: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.348, 95% CI 2-sided [-0.064 to 0.760], Standard Error of Mean 0.2090 — Comparison of FVC, Day 1, 9 hour
Statistical Analysis 44: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.245, 95% CI 2-sided [-0.230 to 0.720], Standard Error of Mean 0.2410 — Comparison of FVC, Day 1, 12 hour
Statistical Analysis 45: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.162, 95% CI 2-sided [-0.245 to 0.569], Standard Error of Mean 0.2063 — Comparison of FVC, Day 1, 24 hour
Statistical Analysis 46: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.535, 95% CI 2-sided [-0.038 to 1.108], Standard Error of Mean 0.2907 — Comparison of FVC, Day 7, Baseline
Statistical Analysis 47: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.623, 95% CI 2-sided [0.072 to 1.175], Standard Error of Mean 0.2798 — Comparison of FVC, Day 7, 1 hour
Statistical Analysis 48: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.459, 95% CI 2-sided [-0.083 to 1.000], Standard Error of Mean 0.2748 — Comparison of FVC, Day 7, 2 hour
Statistical Analysis 49: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.464, 95% CI 2-sided [-0.069 to 0.997], Standard Error of Mean 0.2705 — Comparison of FVC, Day 7, 4 hour
Statistical Analysis 50: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.445, 95% CI 2-sided [-0.104 to 0.994], Standard Error of Mean 0.2786 — Comparison of FVC, Day 7, 9 hour
Statistical Analysis 51: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.284, 95% CI 2-sided [-0.314 to 0.882], Standard Error of Mean 0.3034 — Comparison of FVC, Day 7, 12 hour
Statistical Analysis 52: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.384, 95% CI 2-sided [-0.162 to 0.929], Standard Error of Mean 0.2766 — Comparison of FVC, Day 7, 24 hour

12. Primary Outcome: Number of Participants Who Used Rescue Medication
Description: Inhaled salbutamol was used as a rescue medication. Participants were required to keep a diary of their rescue medication (total number of salbutamol doses taken) over the entire 7-day treatment period. Diaries were reviewed by the Investigator when participants were admitted to the unit on Days 1, 2, 7 and 8.
Time Frame: Up to Day 7
Population: All subject population was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Participants | 0 | 4 | 2

13. Primary Outcome: Number of Participants With Abnormalities in Chemistry Data of Clinical Concern
Description: Clinical chemistry parameters included urea, potassium, aspartate aminotransferase (AST), total bilirubin, creatinine, creatine kinase, chloride, alanine aminotransferase (ALT), uric acid, glucose, gamma glutamyltransferase (GGT), albumin, sodium, phosphorus inorganic, calcium, alkaline phosphatase (ALP) and total protein. It was assessed on Day 1 (pre-dose, 24 hours) and Day 7 (pre-dose, 24 hours). Data for parameters with above and below the potential clinical concern (PCI) is provided.
Time Frame: Up to Day 7
Population: All subject population was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Participants
  Glucose, High | 0 | 1 | 0
  Inorganic phosphorus, Low | 0 | 0 | 1
  Inorganic phosphorus, High | 0 | 0 | 1

14. Primary Outcome: Number of Participants With Abnormalities in Hematology Data of Clinical Concern
Description: Hematology parameters included platelet count, red blood cell (RBC) count, mean corpuscular volume (MCV), total neutrophils, white blood cell (WBC) count (absolute), mean corpuscular hemoglobin (MCH), lymphocytes, mean corpuscular hemoglobin concentration (MCHC), monocytes, hemoglobin, eosinophils, hematocrit and basophils. It was assessed on Day 1 (pre-dose, 24 hours) and Day 7 (pre-dose, 24 hours). Data for parameters with above and below the PCI is provided.
Time Frame: Up to Day 7
Population: All subject population was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Participants | 0 | 0 | 0

15. Primary Outcome: Summary of Microscopy Data for Participants With Abnormal Urinalysis Dipstick Results
Description: Urinalysis parameters included protein, blood, ketones, glucose, bilirubin, urobilinogen, leukocyte esterase, specific gravity, nitrites and pH. Sediment microscopy was performed only on urine samples showing an abnormality on the dipstick. Microscopy was performed for: WBC, RBC, hyaline casts, granular casts and cellular casts. It was assessed on Day 1 (pre-dose, 24 hours) and Day 7 (pre-dose, 24 hours).
Time Frame: Up to Day 7 (pre dose)
Population: All subject population was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Participants
  Urine microscopy-RBC-Day 1 | 1 | 0 | 0
  Urine microscopy-RBC-Day 7 | 1 | 1 | 0
  Urine microscopy-WBC-Day 1 | 0 | 0 | 1
  Urine microscopy-WBC-Day 7 | 1 | 1 | 1

16. Primary Outcome: Summary of Mean (0-24 Hour) and Maximum (0-24 Hour) Heart Rate Measured Using 24 Hour Using Holter ECG Data
Description: Holter monitors were switched on immediately prior to dosing (up to 15mins pre-dose) so as to capture Holter ECG data from the 24 hour period following dosing. It was assessed on Day 1 and 7.
Time Frame: Up to Day 7
Population: All subject population was used.
Measure: Least Squares Mean (95% Confidence Interval); unit: Beats per minute
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 6 | 9 | 8
Beats per minute
  Maximum heart rate, Day 1 | 113.35 [108.13 to 118.57] | 115.58 [111.24 to 119.93] | 112.08 [107.62 to 116.54]
  Maximum heart rate, Day 7 | 114.02 [101.35 to 126.69] | 119.75 [109.21 to 130.30] | 115.01 [104.18 to 125.84]
  Mean heart rate, Day 1 | 71.260 [65.915 to 76.605] | 73.994 [69.498 to 78.491] | 70.186 [65.593 to 74.779]
  Mean heart rate, Day 7 | 68.670 [64.101 to 73.238] | 73.453 [69.610 to 77.295] | 70.239 [63.313 to 74.164]
Statistical Analysis 1: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 2.233, 95% CI 2-sided [-4.743 to 9.210], Standard Error of Mean 3.3333 — Comparison of maximum heart rate Day 1
Statistical Analysis 2: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 5.730, 95% CI 2-sided [-11.200 to 22.664], Standard Error of Mean 8.0907 — Comparison of maximum heart rate Day 7
Statistical Analysis 3: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -1.272, 95% CI 2-sided [-8.051 to 5.507], Standard Error of Mean 3.2390 — Comparison of maximum heart rate Day 1
Statistical Analysis 4: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 0.988, 95% CI 2-sided [-15.470 to 17.443], Standard Error of Mean 7.8616 — Comparison of maximum heart rate Day 7
Statistical Analysis 5: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 2.734, 95% CI 2-sided [-4.468 to 9.936], Standard Error of Mean 3.4410 — Comparison of mean heart rate Day 1
Statistical Analysis 6: Comparison: Placebo vs GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 4.783, 95% CI 2-sided [-1.372 to 10.938], Standard Error of Mean 2.9409 — Comparison of mean heart rate Day 7
Statistical Analysis 7: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = -1.074, 95% CI 2-sided [-8.003 to 5.854], Standard Error of Mean 3.3103 — Comparison of mean heart rate Day 1
Statistical Analysis 8: Comparison: Placebo vs GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Mean Difference (Net) = 1.569, 95% CI 2-sided [-4.353 to 7.490], Standard Error of Mean 2.8291 — Comparison of mean heart rate Day 7

17. Secondary Outcome: Plasma Concentrations of GSK233705
Description: Blood samples were collected at indicated time points. 12 hour pharmacokinetic (PK) sampling was before evening dose.
Time Frame: Day 1 and 7 morning: pre-dose, 5, 15 minutes, 1, 6 and 12 hours post-dose and Day 1 and 7 evening: pre-dose, 5 and 30 post-dose
Population: PK population was used; this was defined as all participants in the all subjects population for whom a PK sample was obtained and analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter
Arm/Group | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 9 | 8
Nanograms per milliliter
  Day 1, AM dose, pre-dose | NA (NA) — NA indicates data not quantifiable. | NA (NA) — NA indicates data not quantifiable.
  Day 1, AM dose, 5 minutes | 0.039 (0.0332) | 0.181 (0.0948)
  Day 1, AM dose, 15 minutes | 0.028 (0.0128) | 0.090 (0.0331)
  Day 1, AM dose, 1 hour | 0.012 (NA) — NA indicates data not quantifiable. | 0.034 (0.0115)
  Day 1, AM dose, 6 hour | NA (NA) — NA indicates data not quantifiable. | NA (NA) — NA indicates data not quantifiable.
  Day 1, AM dose, 12 hour | NA (NA) — NA indicates data not quantifiable. | NA (NA) — NA indicates data not quantifiable.
  Day 1, PM dose, 5 minutes: number analyzed (Participants) | 8 | 8
  Day 1, PM dose, 5 minutes | 0.070 (0.0327) | 0.209 (0.1066)
  Day 1, PM dose, 30 minutes: number analyzed (Participants) | 8 | 8
  Day 1, PM dose, 30 minutes | 0.024 (0.0087) | 0.062 (0.0120)
  Day 7, AM dose, pre-dose: number analyzed (Participants) | 8 | 8
  Day 7, AM dose, pre-dose | 0.013 (0.0111) | 0.024 (0.0070)
  Day 7, AM dose, 5 minutes | 0.062 (0.0513) | 0.226 (0.1257)
  Day 7, AM dose, 15 minutes | 0.046 (0.0291) | 0.146 (0.0724)
  Day 7, AM dose, 1 hour | 0.025 (0.0119) | 0.061 (0.0210)
  Day 7, AM dose, 6 hour | 0.015 (0.0081) | 0.028 (0.0085)
  Day 7, AM dose, 12 hour | NA (NA) — NA indicates data not quantifiable. | 0.028 (0.0242)
  Day 7, PM dose, 5 minutes | 0.068 (0.0477) | 0.218 (0.1091)
  Day 7, PM dose, 30 minutes | 0.028 (0.0115) | 0.064 (0.0233)

18. Secondary Outcome: Urine Concentrations of GSK233705
Description: Urine GSK233705 pharmacokinetic excretion rate-time data is presented. Urine samples were collected throughout study and consolidated data is presented as 0-12 hours and 12-24 hours. 12 hour pharmacokinetic sampling was before evening dose.
Time Frame: Day 1 and 7 throughout 24 hours
Population: PK population was used.
Measure: Mean (Standard Deviation); unit: Nanograms per liter
Arm/Group | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 9 | 8
Nanograms per liter
  Day 1, 0-12 hours | 124.6721 (35.34371) | 348.9206 (110.1697)
  Day 1, 12-24 hours | 179.4939 (47.34615) | 431.8806 (122.7514)
  Day 7, 0-12 hours | 316.6091 (80.41509) | 629.6146 (311.2823)
  Day 7, 12-24 hours | 311.6291 (131.1778) | 643.1492 (218.4276)

19. Secondary Outcome: Derived Plasma PK Parameters-area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUC0-tau)
Description: Blood samples were collected at indicated time points. 12 hour PK sampling was before evening dose. Data presented for morning samples.
Time Frame: as for outcome 17
Population: PK population was used.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour×Nanograms per milliliter
Arm/Group | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 9 | 8
Hour×Nanograms per milliliter
  Day 1: number analyzed (Participants) | 4 | 7
  Day 1 | 0.044 (28.2) | 0.147 (43.0)
  Day 7 | 0.189 (39.3) | 0.430 (44.5)

20. Secondary Outcome: Derived Plasma PK Parameters-area Under Concentration-time Curve From Time 0 to Time of Last Quantifiable Concentration (AUC0-t)
Description: Blood samples were collected at indicated time points. 12 hour PK sampling was before evening dose. Data presented for morning sample as adjusted geometric mean.
Time Frame: as for outcome 17
Population: PK population was used.
Measure: Geometric Mean (90% Confidence Interval); unit: Hour×Nanograms per milliliter
Arm/Group | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 9 | 8
Hour×Nanograms per milliliter
  Day 1 | 0.016 [0.011 to 0.021] | 0.053 [0.038 to 0.073]
  Day 7 | 0.018 [0.013 to 0.025] | 0.056 [0.039 to 0.080]
Statistical Analysis 1: Comparison: GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Ratio = 1.139, 90% CI 2-sided [0.811 to 1.601], Standard Error of Mean 0.1939 — SE logs is presented as standard error of mean. Comparison of GSK233705 50 µg twice daily Day 7 versus Day 1
Statistical Analysis 2: Comparison: GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Ratio = 1.060, 90% CI 2-sided [0.739 to 1.520], Standard Error of Mean 0.2057 — SE logs is presented as standard error of mean. Comparison of GSK233705 100 µg twice daily Day 7 versus Day 1

21. Secondary Outcome: Derived PK Plasma Parameters-area Under Concentration-maximum Observed Plasma Concentration (Cmax)
Description: Blood samples were collected at indicated time points. 12 hour PK sampling was before evening dose. Data presented for morning and evening samples as adjusted geometric mean.
Time Frame: as for outcome 17
Population: PK population was used.
Measure: Geometric Mean (90% Confidence Interval); unit: Nanograms per liter
Arm/Group | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 9 | 8
Nanograms per liter
  AM Dose, Day 1 | 0.035 [0.025 to 0.050] | 0.160 [0.109 to 0.234]
  AM Dose, Day 7 | 0.049 [0.031 to 0.078] | 0.190 [0.117 to 0.309]
  PM Dose, Day 1 | 0.052 [0.035 to 0.077] | 0.186 [0.123 to 0.281]
  PM Dose, Day 7 | 0.051 [0.032 to 0.080] | 0.191 [0.119 to 0.309]
Statistical Analysis 1: Comparison: GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Ratio = 1.408, 90% CI 2-sided [0.934 to 2.122], Standard Error of Mean 0.2340 — SE logs is presented as standard error of mean. Comparison of Cmax AM dose for GSK233705 50 µg twice daily Day 7 versus Day 1
Statistical Analysis 2: Comparison: GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Ratio = 1.190, 90% CI 2-sided [0.770 to 1.838], Standard Error of Mean 0.2482 — SE logs is presented as standard error of mean. Comparison of Cmax AM dose for GSK233705 100 µg twice daily Day 7 versus Day 1
Statistical Analysis 3: Comparison: GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Ratio = 0.979, 90% CI 2-sided [0.658 to 1.457], Standard Error of Mean 0.2269 — SE logs is presented as standard error of mean. Comparison of Cmax PM dose for GSK233705 50 µg twice daily Day 7 versus Day 1
Statistical Analysis 4: Comparison: GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Ratio = 1.028, 90% CI 2-sided [0.674 to 1.568], Standard Error of Mean 0.2407 — SE logs is presented as standard error of mean. Comparison of Cmax PM dose for GSK233705 100 µg twice daily Day 7 versus Day 1

22. Secondary Outcome: Derived PK Plasma Parameters-area Under Concentration-time of Maximum Observed Plasma Concentration (T-max), Half-life (T-half) and Last Time Point Where the Concentration is Above the Limit of Quantification (T-last)
Description: Blood samples were collected at indicated time points. 12 hour PK sampling was before evening dose. Data presented for morning and evening samples.
Time Frame: as for outcome 17
Population: PK population was used.
Measure: Median (Full Range); unit: Hour
Arm/Group | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 9 | 8
Hour
  T-half, Day 1, AM dose: number analyzed (Participants) | 4 | 7
  T-half, Day 1, AM dose | 0.624 [0.50 to 1.08] | 1.167 [0.71 to 2.25]
  T-half, Day 7, AM dose: number analyzed (Participants) | 5 | 5
  T-half, Day 7, AM dose | 4.122 [1.66 to 7.01] | 7.189 [6.59 to 13.97]
  T-last, Day 1, AM dose | 1.000 [0.48 to 2.00] | 2.025 [2.00 to 6.00]
  T-last, Day 7, AM dose | 11.920 [2.00 to 12.03] | 11.920 [11.92 to 12.08]
  T-last, Day 1, PM dose | 0.500 [0.25 to 0.50] | 0.500 [0.48 to 0.52]
  T-last, Day 7, PM dose | 0.500 [0.48 to 0.53] | 0.500 [0.50 to 0.53]
  T-max, Day 1, AM dose | 0.080 [0.08 to 1.98] | 0.080 [0.08 to 0.10]
  T-max, Day 7, AM dose | 0.230 [0.08 to 6.00] | 0.080 [0.08 to 0.10]
  T-max, Day 1, PM dose | 0.080 [0.08 to 0.47] | 0.080 [0.08 to 0.10]
  T-max, Day 7, PM dose | 0.080 [0.08 to 0.48] | 0.080 [0.08 to 0.12]

23. Secondary Outcome: Derived Urine Pharmacokinetic (PK) Parameters-area Under the Plasma Concentration-amount of Drug Excreted Unchanged in Urine (Ae)
Description: Urine GSK233705 pharmacokinetic excretion rate-time data is presented. Urine samples were collected throughout study and consolidated data presented as AM dose and PM dose. 12 hour pharmacokinetic sampling was before evening dose.
Time Frame: Day 1 and 7 throughout 24 hours
Population: PK population was used.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram
Arm/Group | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 9 | 8
Nanogram
  Ae, Day 1, AM dose | 1432.6 (30.6) | 3977.1 (32.4)
  Ae, Day 7, AM dose | 3661.2 (27.4) | 6538.3 (66.5)
  Ae, Day 1, PM dose | 2080.2 (29.5) | 4913.3 (39.0)
  Ae, Day 7, PM dose | 3344.7 (62.0) | 7328.5 (36.6)
Statistical Analysis 1: Comparison: GSK233705 50 µg Twice Daily; Test type: Superiority or Other; Ratio = 2.556, 90% CI 2-sided [2.033 to 3.213], Standard Error of Mean 0.131 — SE logs is presented as standard error of mean. Comparison of Ae AM dose for GSK233705 50 µg twice daily Day 7 versus Day 1
Statistical Analysis 2: Comparison: GSK233705 100 µg Twice Daily; Test type: Superiority or Other; Ratio = 1.644, 90% CI 2-sided [1.290 to 2.095], Standard Error of Mean 0.138 — SE logs is presented as standard error of mean. Comparison of Ae AM dose for GSK233705 100 µg twice daily Day 7 versus Day 1

24. Secondary Outcome: Derived Urine PK Parameters-area Under Concentration-fraction of Dose Excreted Unchanged in Urine (Fe)
Description: Urine GSK233705 pharmacokinetic excretion rate-time data is presented. Urine samples were collected throughout study and consolidated data presented as 0-12 hours and 12-24 hours. 12 hour pharmacokinetic sampling was before evening dose.
Time Frame: Day 1 and 7 throughout 24 hours
Population: PK population was used.
Measure: Mean (Standard Deviation); unit: Percentage of dose
Arm/Group | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 9 | 8
Percentage of dose
  Day 1, AM dose | 3.0 (0.84) | 4.2 (1.30)
  Day 7, AM dose | 7.5 (1.88) | 7.5 (3.67)
  Day 1, PM dose | 4.3 (1.14) | 5.2 (1.48)
  Day 7, PM dose | 7.5 (3.15) | 7.7 (2.66)

25. Secondary Outcome: Derived Urine PK Parameters-area Under Concentration-renal Clearance (Clr)
Description: Urine GSK233705 pharmacokinetic excretion rate-time data is presented. Urine samples were collected throughout study. 12 hour pharmacokinetic sampling was before evening dose.
Time Frame: Day 1 and 7 throughout 24 hours
Population: PK population was used. Only those participants available at the specified time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
Number analyzed (Participants) | 9 | 8
Liters per hour
  Day 1: number analyzed (Participants) | 4 | 7
  Day 1 | 36.2 (24.5) | 27.5 (50.2)
  Day 7 | 19.4 (49.1) | 15.2 (68.4)

ADVERSE EVENTS:
Time Frame: All AE and SAE were reported until he or she has completed the study (including any follow-up period). This included 28 days of screening and 17 days of treatment and follow-up (approximately 45).
Description: All subjects population was used for reporting non-SAE and SAE.
Arm/Group | Placebo | GSK233705 50 µg Twice Daily | GSK233705 100 µg Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 4/6 | 4/9 | 4/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | GSK233705 50 µg Twice Daily (N=9) | GSK233705 100 µg Twice Daily (N=8)
Fatigue (General disorders) | 1 | 1 | 1
Catheter site related reaction (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Infusion site irritation (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2
Somnolence (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.